CLINICAL TRIAL: NCT05829772
Title: Community-based Monitoring of Cholera Antibodies' Seroprevalence, and Home Follow-up of Positive Cases, in the Context of Cholera Vaccination Campaign, Democratic Republic of the Congo
Brief Title: Impact Study of Cholera Vaccination in Endemic Areas - Seroprevalence
Status: Completed | Type: Observational
Sponsor: Epicentre (Other)
Collaborators: Wellcome Trust (Other); Institut Pasteur (Industry); Institut National de Recherche Biomédicale. Goma, République Démocratique du Congo (Unknown); Ministry of Public Health, Democratic Republic of the Congo (Other Government); Medecins Sans Frontieres, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2146-WT
Record Dates: First submitted 2023-04-13; First posted 2023-04-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cholera
Keywords: Cholera incidence rates; Mass vaccination campaign; V.Cholerae; Serial seroprevalence
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Full blood serum samples are collected for all participants in each surveys, 4 in Goma and 3 in Bukama. An additional EDTA tube is also collected in 2 surveys (1st in Goma and 1st in Bukama). They will be analyzed for cholera antibody levels (Luminex and/or vibriocidal assay). In addition, stool samples will be collected in 1 survey in Goma and RDT-tested. Participants with positive samples will be proposed to participate in home follow-up study. During home follow-up, a stool sample will be collected from all household members upon household visits.On day 90and180, stool samples will only be collected from participants who tested positive for cholera shedding during the previous visits.Samples from peri-household environment (drinking water, kitchen swab, latrine swab and latrine sludge), will be taken during the first 3 household visits and sent to laboratory.Environment samples collection will be stopped afterwards if all of them tested negative for at least 2 consecutive visits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This project aims to fill this essential knowledge gap by assessing the impact of oral cholera vaccine mass campaigns in 2 sites (urban and rural) in DRC, described in this protocol. The evidence generated from this project will be key to develop future strategies regarding cholera vaccine use in endemic settings, including places with higher burden in terms of cholera mortality

DETAILED DESCRIPTION:
The project will comprise three different components:

Clinical cholera surveillance to measure cholera diseases incidence in selected African hotspots targeted by vaccination.

Serial serological surveys to measure the prevalence of recent cholera infection (within the last 12 months).

Identification and follow up of individuals with positive V. cholerae shedding (symptomatic or asymptomatic) among sero-survey participants and among household members of cholera confirmed cases.

The present protocol relates to the setup of seroprevalence surveys and the follow up of individuals with positive V. cholerae shedding identified through seroprevalence surveys, in DRC.

This protocol will allow us to assess if a large vaccination campaign reaching high coverage in cholera hotspot in Africa can allow sustained control of cholera for at least two years, by fulfilling the following specific objectives:

1. To calculate the proportion of individuals infected with cholera recently (i.e. previous year or last 2 months) before the campaign distribution or in non-vaccinated zones (baseline survey, rural site) or following the mass OCV campaign and before the start of the usual cholera season (pre-season survey, urban site).
2. To assess proportion of individuals recently infected (i.e. infected in the last two months or in the last year) during the expected peak-week of cholera in the area (peak survey, urban site) and at the end of the expected cholera season (post-season survey), as compared to baseline or pre-season survey.
3. To assess the intra-household transmission and correlation in cholera recent infections among vaccinated and non-vaccinated households (post-season survey)
4. To compare mortality linked to diarrheal diseases and potential cholera in the community of rural site before and after vaccination
5. To assess the duration of shedding among vaccinated and unvaccinated individuals and the duration of viable V. cholerae in the peri-household environment.
6. To measure the secondary cholera attack rates (symptomatic and asymptomatic) at household level among vaccinated and unvaccinated individuals following the identification of an index case in a given household.

ELIGIBILITY:
Inclusion Criteria:

* All persons,

  1. Living in the randomly-selected households in targeted area AND
  2. Randomly selected among household members. Inclusions will be limited to 1 participant per household, except for one survey AND
  3. Giving his/her consent (or assent for children 13 to 17 years old) to participate in the study

Exclusion Criteria:

* People who decline to participate will be excluded from the study. For 2nd survey in Goma only: members of the household who cannot be reached after 2 attempts will be excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants are selected randomly in the community. GPS point selection is made on mapping of roofs from the area, and some roofs are randomly selected with appropriate GIS software. Persons living under the randomly selected roof are proposed to participate in the surveys, or close neighboors in case of refusal.
Sampling Method: Non-Probability Sample
Enrollment: 7000 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
To better characterize cholera immunization in the population of cholera hotspot in Africa and assess the impact of a large vaccination campaign reaching high coverage | 2 years
  Cholera-specific antibody levels will be measured in all participants for each surveys. Serial surveys will allow monitoring level of antibodies over time following the vaccination campaign

SECONDARY OUTCOMES:
Calculate proportion of individuals infected with cholera (previous year or last 2 months) before the campaign distribution or in non-vaccinated zones or following the massOCV campaign and before the start of cholera season:pre-season survey, urban site. | 2 years
Assess proportion of individuals infected (the last 2 months or previous year) during the expected peak-week of cholera in the area and at the end of the expected cholera season (post-season survey), as compared to baseline or pre-season survey. | 2years
To assess the intra-household transmission and correlation in cholera recent infections among vaccinated and non-vaccinated households (post-season survey) | 2 years
To compare mortality linked to diarrheal diseases and potential cholera in the community of rural site before and after vaccination | 2 years
To assess the duration of shedding among vaccinated and unvaccinated individuals and the duration of viable V. cholerae in the peri-household environment. | 2 years
To measure the secondary cholera attack rates (symptomatic and asymptomatic) at household level among vaccinated and unvaccinated individuals following the identification of an index case in a given household. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia Porten, Study Director — Epicentre; Francisco Luquero, Study Chair — Gavi
Locations (2):
- Democratic Republic of the Congo (2):
  - Epicentre/Médecins Sans Frontières, Bukama, Haut-Lomami
  - Médecins Sans Frontières France, Goma, North Kivu

IPD SHARING:
Plan to Share IPD: No